CLINICAL TRIAL: NCT06070389
Title: Polysomnography Validation of the Sansa Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huxley Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EDS-50031
Record Dates: First submitted 2023-06-16; First posted 2023-10-06 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Sleep-Disordered Breathing
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Sansa device — The Sansa device will be used during a single overnight polysomnography study.

SUMMARY:
The objective of this study is to evaluate the performance of the Sansa device for the diagnosis of sleep disordered breathing.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* able to read, understand, and sign informed consent documentation
* willing to sleep with the Sansa device and PSG simultaneously in the sleep clinic
* suspected or known to have sleep disordered breathing

Exclusion Criteria:

* exhibit deformities of the chest that would interfere with sensor placement
* have broken or injured skin that would interfere with sensor placement
* known to experience adverse reactions to medical-grade adhesive
* diagnosed with hypoventilation
* diagnosed with severe chronic obstructive pulmonary disease
* exhibit symptoms of significant non-respiratory sleep disorders
* diagnosed with a neuromuscular disorder leading to muscle weakness
* chronically use supplemental oxygen at night or during the day
* pregnant
* scheduled to undergo titration of a hypoglossal nerve stimulation device
* undergo permanent pacing with an implanted pacemaker
* diagnosed with congestive heart failure with an ejection fraction less than 45%

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 533 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2023-12-13 (Actual)

PRIMARY OUTCOMES:
Sensitivity and Specificity of the Sansa device to detect sleep disordered breathing compared to polysomnography | 1 night

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Goldstein, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - Pulmonary & Sleep Specialists, Decatur, Georgia
  - University of Michigan, Ann Arbor, Michigan

REFERENCES:
- [Derived] Goldstein C, Ghanbari H, Sharma S, Collop N, Namen A, Kirsch DB, Drucker M, Khayat R, Pollock M, Torstrick B, Walsh C, Herreshoff E, Frankel DS, Rosen IM. Polysomnography validation of SANSA to detect obstructive sleep apnea. Front Neurol. 2025 Jun 16;16:1592690. doi: 10.3389/fneur.2025.1592690. eCollection 2025. PMID 40589991